CLINICAL TRIAL: NCT04863963
Title: Milligan-Morgan Hemorrhoidectomy Versus Dearterialization With Mucopexy in the Treatment of Grade III Hemorrhoidal Disease: Multicenter Retrospective Study
Brief Title: Milligan-Morgan Versus Dearterialization With Mucopexy
Acronym: EMODART3
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Aquila (Other)
Responsible Party: Principal Investigator, Lucia Romano, Principal Investigator, Università degli Studi dell'Aquila
Other Study IDs: Observational
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hemorrhoids; Hemorrhoid Prolapse
Keywords: Hemorrhoids; Milligan- Morgan; Mucopexy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Milligan Morgan: Patients aged ≥18 years-old, with Goligher's grade III haemorrhoidal disease, who underwent elective Milligan-Morgan hemorrhoidectomy surgery.
  Interventions: Procedure: Milligan Morgan
- Dearterialization with mucopexy: Patients aged ≥18 years-old, with Goligher's grade III haemorrhoidal disease, who underwent elective Doppler-guided or non-Doppler guided HAL surgery associated with mucopexy

INTERVENTIONS:
Procedure: Milligan Morgan — Surgical intervention used in case of Goligher's grade III hemorrhoidal disease
  Other Names: Transanal dearterialization with mucopexy
  Groups: Milligan Morgan

SUMMARY:
Nowadays, there are several methods that can be used for grade III hemorrhoidal disease, according to Goligher classificiation. Milligan Morgan hemorrhoidectomy is considered the most effective treatment in many centers, even if characterized by marked postoperative pain. Among the minimally invasive alternative procedures, the transanal hemorrhoidal dearterialization (HAL - ligation of the hemorrhoidal artery) Doppler-guided or without Doppler, associated with mucopexy, seems to gain success, with promising results but still awaiting high-grade scientific evidence.

On the basis of this background, we decided to carry out a multi-center survey on a national scale, retrospectively including patients diagnosed with Goligher's grade III hemorrhoidal disease, surgically treated with hemorrhoidectomy or dearterialization.

DETAILED DESCRIPTION:
The study will be of a multicentre observational retrospective type. Any Italian Center belonging to the Italian Society of Colorectal Surgery (SICCR) in which at least 30 procedures are performed per year for haemorrhoidal disease can join the study. Each Center must identify a Head of the study and a maximum of 2 collaborators. Each Center participating in the Study will be provided with a data collection sheet for completion. The information regarding the follow-up may come from a telephone survey or an outpatient clinical visit. In both cases, the patient will be asked to express informed consent by filling in the form attached to the information sheet.

The study will include patients treated with the analysed methods (Milligan Morgan or hemorrhoidal dearterialization) in the period comprising the 4 years prior to the adhesion of the center to the survey.

Patients included in the study will need to have at least 24 months of follow-up.

Given the inevitable effects of the SARS-CoV-2 pandemic on surgical and outpatient activities, the study period is considered valid until February 2020. Data regarding surgery or follow-up after March 2020 will not be included in analyzes.

The participation of 435 patients for each group is expected (870 total patients) considering a power of 80%, of which at least 50 in this facility, over the age of 18.

Clinical recovery is defined as the disappearance of the proctological symptoms reported by the patient (post-operative symptom score equal to 0).

Instead, anatomical healing is defined as the absence of haemorrhoidal pathology on objective examination (maximum Gholigher's grade 1).

Relapse is defined as the persistence or reappearance of the reported symptoms and the finding on physical examination of hemorrhoidal disease of a degree equal to or higher than the assessment attributed during the preoperative examination.

The physical examination is conducted by the same medical staff who made the diagnosis.

Symptoms will be assessed using the symptom score system proposed by Giordano et al., according to which the patient is asked to assign a score to each parameter evaluated, ranging from 0 (absence of symptoms) to 4 (daily symptoms or at each evacuation). The parameters evaluated are bleeding, prolapse, the need for manual reduction, pain or discomfort and the impact on quality of life. An overall score of 0 corresponds to the total absence of symptoms, while an overall score of 20 indicates the worst possible symptomatology.

The patient will be asked to assign a score to the symptoms present before the surgery and therefore 24 months after the same.

According to the data in the literature, the following factors could be associated with a higher risk of relapse: female sex, presence of associated mucosal prolapse.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years-old
* Goligher's grade III haemorrhoidal disease
* indication to elective Doppler-guided or non-Doppler guided HAL surgery associated with mucopexy or Milligan-Morgan hemorrhoidectomy.

Exclusion Criteria:

* Recurrent disease
* bleeding disorders
* chronic inflammatory bowel diseases
* vasculopathies
* combined surgical techniques (HAL with mucopexy and removal of one or more haemorrhoidal nodules)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be of a multicentre observational retrospective type. Any Italian Center belonging to the Italian Society of Colorectal Surgery (SICCR) in which at least 30 procedures are performed per year for haemorrhoidal disease can participate.
  The study will include patients treated with the aforementioned methods in the period including the 4 years prior to the adhesion of the center to the survey.
  All patients aged ≥18 years-old, with Goligher's grade III haemorrhoidal disease can be included in the study, who underwent elective Doppler-guided or non-Doppler guided HAL surgery associated with mucopexy or Milligan-Morgan hemorrhoidectomy.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Rate of complications | 24 months
  Compare surgical techniques in terms of complications
Effectiveness | 24 months
  Compare surgical techniques in terms of effectiveness (persistence / reappearance of symptoms and recurrences).
Speed in functional recovery | 24 months
  Compare surgical techniques in terms of functional recovery
Rate of choice of the two techniques | 24 months
  Evaluate the rate of choice in Italy of the two different surgical techniques (HAL THD with mucopexy and Milligan Morgan hemorrhoidectomy) for the treatment of Golighers's grade III hemorrhoidal disease

SECONDARY OUTCOMES:
Surgical device | 24 months
  Analyze the surgical devices used
Type of anesthesia | 24 months
  Evaluate the type of anesthesia choiced
Hospitalization times | 24 months
  Evaluate and compare hospitalization times

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Giuliani, L’Aquila, AQ, Italy

REFERENCES:
- [Derived] Giuliani A, Romano L, Necozione S, Cofini V, Di Donato G, Schietroma M, Carlei F; EMODART3 Study Group. Excisional Hemorrhoidectomy Versus Dearterialization With Mucopexy for the Treatment of Grade III Hemorrhoidal Disease: The EMODART3 Multicenter Study. Dis Colon Rectum. 2023 Dec 1;66(12):e1254-e1263. doi: 10.1097/DCR.0000000000002885. Epub 2023 Aug 24. PMID 37616177